CLINICAL TRIAL: NCT01264328
Title: "Phase II Study of the Combination of Panitumumab With Paclitaxel as First-line Treatment of Subjects With Metastatic or Recurrent Head and Neck Cancer"
Brief Title: Study of the Combination of Panitumumab With Paclitaxel as First-line Treatment of Subjects With Head and Neck Cancer
Acronym: VECTITAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (Other)
Collaborators: Amgen (Industry); Trial Form Support S.L. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTCC-2009-03
Record Dates: First submitted 2010-12-02; First posted 2010-12-21 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer, panitumumab, TTCC-2009-03
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Panitumumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab + Paclitaxel (Experimental): Treatment consisted of intravenous panitumumab 6 mg/kg q2w, administered in one hour the first day and in 30 minutes thereafter (if no infusional reaction was observed) plus intravenous paclitaxel 80 mg/m2 weekly administered one hour after panitumumab in one hour infusion, until progression or unacceptable toxicity. Panitumumab does not require prophylactic premedication from the first infusion. Paclitaxel was administered with: dexamethasone 10 mg, diphenhydramine 30 mg and antiH2 (cimetidine 300 mg or ranitidine 50 mg). Dose modifications of paclitaxel included 4.8 mg/kg (80% of the initial dose) and 3.6 mg/kg (60%) when recovered from a grade 3-4 skin toxicity to grade ≤2. Continuing paclitaxel on the day of the planned infusion required no grade ≥2 mucositis and hematologic recovery with an absolute neutrophil count ≥1,500/ml and a platelet count ≥75,000.
  Interventions: Drug: Panitumumab + paclitaxel

INTERVENTIONS:
Drug: Panitumumab + paclitaxel — Paclitaxel 80 mg/m2 may be infused, intravenously, over one hour every week. Panitumumab will be administered every 2 weeks at a dose of 6 mg/kg, using a non pyrogenic low protein binding filter with a 0.20-0.22-μm pore size intravenously over 1 hour ± 15 minutes. Panitumumab will be administered prior to paclitaxel.
  Other Names: Vectibix®

SUMMARY:
The clinical hypothesis of this study is that the first-line treatment with the combination of panitumumab and paclitaxel will provide benefit for patients with metastatic or current Squamous Cell Carcinoma of the Head and Neck (SCCHN)

DETAILED DESCRIPTION:
Panitumumab, a fully human IgG2 anti-EGFR monoclonal antibody, has shown activity in preclinical models of SCCHN, and promising activity in refractory SCCHN patients in a phase I clinical trial. Recently, the investigators also reported encouraging outcomes of anti-EGFR-paclitaxel combination in a phase II study. On the basis of this background, a phase II clinical trial (VECTITAX study) was designed with the objective of evaluating the activity and safety profile of panitumumab in combination with paclitaxel in patients with recurrent or metastatic SCCHN.

The VECTITAX study was a single arm, open label, multicenter, phase II clinical trial. To be included patients had to have histologically or cytologically confirmed SCCHN. The current situation had to be recurrent or metastatic, deemed to be untreatable by surgery or radiotherapy. No previous systemic antineoplastic therapy for the recurrent/metastatic disease may have been administered. However, previous chemotherapy was allowed as a part of a multimodality radical treatment if completed >24 weeks before study entry.

Primary endpoint was confirmed objective response rate (ORR) according to RECIST 1.1 criteria in the intention-to-treat population (ITT). Tumor assessments were planned to be performed every two months. Response confirmation was to be assessed not before 4 weeks after a partial or complete response, or before 6 weeks after a stable disease. Secondary endpoints were disease control rate, time to response, duration of response, progression-free survival (PFS), OS, safety profile and QoL through EQ-5D-3L with visual analogic scale (VAS). Quality of life scores were registered at baseline and every eight weeks thereafter.

Treatment consisted of intravenous panitumumab 6 mg/kg q2w, administered in one hour the first day and in 30 minutes thereafter (if no infusional reaction was observed) plus intravenous paclitaxel 80 mg/m2 weekly administered one hour after panitumumab in one hour infusion, until progression or unacceptable toxicity. Panitumumab does not require prophylactic premedication from the first infusion.

ELIGIBILITY:
Inclusion Criteria:

* Signed Inform Consent
* Age > 18 years
* Histologically or cytologically confirmed SCCHN
* Diagnosis of metastatic disease by the investigator and/or recurrent disease determined to be incurable by surgery or radiotherapy
* Subjects who have received radiation as primary therapy are eligible if radiation therapy treatment was completed > 4 weeks prior to inclusion
* Subjects who have previously received chemotherapy as part of the initial multimodality treatment for locally advanced disease are eligible if the chemotherapy was completed > 24 weeks prior to inclusion
* At least 1 unidimensionally measurable lesion of ≥ 20 mm using conventional techniques or ≥10 mm with spiral CT scan. Target lesions must not be chosen from a previously irradiated field unless there had been documented tumour progression in that lesion prior to inclusion
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1 at screening
* Haematological function:

  * ANC ≥ 1.5 x 109 cells/L
  * Hemoglobin ≥ 9.0 g/dL
  * Platelet count ≥ 100 x 109/L
* Kidney function:

  o Adequate renal function with creatinine clearance ≥ 60 mL/min)
* Liver function:

  * AST ≤ 3 x ULN (if liver metastases, ≤ 5 x ULN)
  * ALT ≤ 3 x ULN (if liver metastases, ≤ 5 x ULN)
  * Bilirubin ≤ 2 x ULN
* Metabolic function:

  * Magnesium ≥ lower limit of normal,
  * Calcium ≥ lower limit of normal

Exclusion Criteria:

* Documented or symptomatic central nervous system metastases
* Nasopharyngeal carcinoma
* History of interstitial lung disease (eg, pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest scan
* History of another primary cancer, except:

  * Curatively treated in situ cervical cancer, or
  * Curatively resected non-melanoma skin cancer or
  * Other primary solid tumour curatively treated with no known active disease present and no treatment administered for ≥ 3 years prior to starting the study treatment. In that case confirmation of inclusion by the sponsor is required.
* Clinically significant cardiovascular disease ≤ 1 year prior to starting the study treatment
* Pulmonary embolism, deep vein thrombosis, or other significant thromboembolic event ≤ 8 weeks prior to starting the study treatment
* Symptomatic peripheral neuropathy of Grade ≥ 2 based on the CTCAE v3.0
* Subjects not recovered from all previous acute radiotherapy-related toxicities to ≤ grade 1
* History of severe skin disorder that in the opinion of the investigator may interfere with study conduct
* Known positive test for human immunodeficiency virus (HIV) infection, hepatitis C virus, acute or chronic hepatitis B infection
* Active infection requiring systemic treatment or any uncontrolled infection ≤ 14 days prior to starting the study treatment
* History of interstitial pneumonia or pulmonary fibrosis or signs of interstitial pneumonia or pulmonary fibrosis on the baseline chest X-ray.
* Known allergy or hypersensitivity to panitumumab, or other study medications.
* Prior anti epidermal growth factor receptor (EGFr) antibody therapy or treatment with small molecule EGFr inhibitors unless received as part of prior multimodality treatment and completed > 24 weeks prior to starting the study treatment. In this case, the investigator should confirm that the subject had not presented any previous cetuximab-related infusion reaction > grade 2.
* Subject is currently enrolled in or ≤ 30 days since ending other investigational device, investigational procedure, or drug study(s), or subject is receiving other investigational agent(s)
* Subjects requiring use of immunosuppressive agents, however, corticosteroids are allowed
* Man or woman of child-bearing potential who do not consent to use adequate contraceptive precautions during the course of the study, and for 6 months after the last study drug administration for women, and 3 months for men.
* Female subject who is pregnant or breast-feeding, or planning to become pregnant within 6 months after the end of treatment.
* Major surgery requiring general anesthesia/ spinal anesthesia and a significant incision ≤ 28 days or minor surgery ≤ 14 days prior to starting the study treatment. Subjects must have recovered from surgery-related toxicities.
* Subjects who do not wish to meet the study requirements or are unable to do so.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03-09 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2014-09-29 (Actual)

PRIMARY OUTCOMES:
objective response rate | 2 years
  To assess the effect of the combination of panitumumab and paclitaxel on objective response rate in first-line treatment of metastatic or recurrent squamous cell carcinoma of head and neck (SCCHN).

SECONDARY OUTCOMES:
Time to response, duration of response, progression free-survival, overall survival. | 2 years
  Secondary Objectives
  * To assess the disease control rate, time to response, duration of response, progression free-survival and overall survival.
  * To estimate changes in patient-reported outcomes (PRO).
  * To describe the safety profile of the combination of panitumumab and paclitaxel.
  1.3 Exploratory Objectives:
  * To investigate the effects of genetic variation in cancer genes and drug target genes on subject response to panitumumab and Paclitaxel combination chemotherapy.
  * To investigate the predictive potential of different biomarkers on efficacy and/or safety endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Jesús Cruz Hernández, Professor, Study Director — University of Salamanca; Javier Martínez Trufero, MD, Principal Investigator — Hospital Miguel Servet de Zaragoza; Juan José Grau, MD, Principal Investigator — Hospital Clínic i Provincial de Barcelona; Joaquina Martínez, MD, Principal Investigator — Hospital Virgen de las Nieves (Granada); Antonio López Pousa, MD, Principal Investigator — Hospital de la Santa Creu i Sant Pau de Barcelona; Alfonso Berrocal, MD, Principal Investigator — Hospital General Universitario de Valencia; Ricardo Hitt, MD, Principal Investigator — Hospital 12 de Octubre de Madrid; Ricardo Mesia, MD, Principal Investigator — Institut Català d'Oncología. Hospital Duran i Reynals de Barcelona; Elvira del Barco Morillo, MD, Study Director — University of Salamanca; Carlos García, MD, Principal Investigator — Hospital General Yagüe de Burgos; Alicia Hurtado, MD, Principal Investigator — Fundación Hospitalaria de Alcorcón de Madrid; Miguel Pastor, MD, Principal Investigator — Hospital La Fe de Valencia; Ruth Vera García, MD, Principal Investigator — Hospital de Navarra
Locations (12):
- Spain (12):
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General de Yagüe, Burgos
  - H. Virgen de las Nieves, Granada
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital General Universitario, Valencia
  - Hospital Universitario la Fe de Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Del Barco Morillo E, Mesia R, Adansa Klain JC, Vazquez Fernandez S, Martinez-Galan J, Pastor Borgonon M, Gonzalez-Rivas C, Caballero Daroqui J, Berrocal A, Martinez-Trufero J, Vera R, Cruz-Hernandez JJ; Spanish Head And Neck Cancer Cooperative Group (TTCC). Phase II study of panitumumab and paclitaxel as first-line treatment in recurrent or metastatic head and neck cancer. TTCC-2009-03/VECTITAX study. Oral Oncol. 2016 Nov;62:54-59. doi: 10.1016/j.oraloncology.2016.09.009. Epub 2016 Oct 8. PMID 27865372
- See also: This site would like to expose the activities of the group and at the same time serve as an information and communication tool of this pathology for professionals and patients. — http://www.ttccgrupo.org